CLINICAL TRIAL: NCT06790459
Title: Effects of Transmucosal Electrical Tongue Stimulation (TUD) on Tonic Pupil Size in the Dark
Brief Title: Effects of the Ultra-low Frequencies TENS on the Arousal Circuits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Sara Di Nicolantonio, PhD candidate, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of L'Aquila
Record Dates: First submitted 2025-01-16; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Pupil Diameter; Arousal
Keywords: Pupil size; ULFTENS; Trigeminal electrical stimulation; tongue stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 20 women of 20-30 years would be enrolled to the experimental group. They will undergone to tongue stimulation with ULFTENS device for 15 minutes. Pupils' diameter will be measure for three time points, before, during and after the tongue stimulation
  Interventions: Device: UlfTens (Ultra-low-frequencies Transcutaneous electrical nervous stimulation)
- Control group (No Intervention): 20 women of 20-30 years will be enrolled to the control group. Their pupils' diameter will be measure at three time points

INTERVENTIONS:
Device: UlfTens (Ultra-low-frequencies Transcutaneous electrical nervous stimulation) — ULFTENS device will be administered in the experimental group for 15 minutes
  Arms: Experimental group

SUMMARY:
Pupil size is associated with the activity of the noradrenergic system, with an increase reflecting a higher state of arousal. Transmucosal electrical stimulation of the tongue could treat disorders related to dysfunctions of this system, and trigeminal stimulation through ULFTENS (TUD) has shown some positive effects. However, no studies have examined the effect of stimulation of the anterior mucosa of the tongue on pupil size as an indicator of arousal. The aim of this study will be to evaluate the effect of ULFTENS stimulation on pupil size in the dark.

DETAILED DESCRIPTION:
Changes in pupil size are indicative of the activity of the noradrenergic system, with pupil dilation associated with a higher state of arousal. According to various studies, odontological ULFTENS, through trigeminal stimulation, can help rebalance this altered system with positive effects. Our goal is to harness the capabilities of ULFTENS by stimulating the dorsal lingual mucosa and evaluating its effects on pupil size in the dark. Healthy women aged between 20 and 30 will be recruited and divided into two groups: a control group and an experimental group. Participants in the control group will lie down on a bed with their eyes closed, and will then be asked to open their eyes without moving their eyelids. Pupil diameter will be measured using a pupillometer for 15 seconds. This procedure will be repeated twice. The experimental group will receive a tongue stimulator connected to the ULFTENS, which will be activated after the first measurement. The stimulation will last approximately 15 minutes, with a second measurement taken after 15 seconds. At the end of the stimulation, the final measurement will be taken. The goal is to measure the pupil diameter of both eyes at the three time points and compare the results between the two groups to assess the effect of the stimulator on arousal circuits.

ELIGIBILITY:
Inclusion Criteria:

* good health status and physical fitness
* female sex
* age between 20 and 30 years
* non-smoker
* no more than 3 espresso coffees per day
* no intake of stimulant or psychotropic drugs in general
* body mass index between 18.5 and 24.9

Exclusion Criteria:

* presence of acute and/or chronic cardiocirculatory and respiratory disorders
* metabolic and autonomic system disorders
* intake of peripheral and central nervous system excitatory or inhibiting substances
* presence of generalized anxiety and/or panic attacks, or mood disorders.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Pupil size | 12 minutes
  left and right pupils diameter will be measured using a pupillometry. Images of the pupils will be acquired by the Oculus system, using two infrared CCD cameras (resolution 720 × 576 pixels, 256 grey levels) mounted on a light helmet (1.5 kg), with sampling frequency of 25 frame/s. The eyes will be illuminated with an infrared diode with 880 nm of wave length.

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Monaco, Principal Investigator — University of L'Aquila
Locations (1):
- Dental Clinic, Mesva department, L’Aquila, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monaco A, Cattaneo R, Smurra P, Di Nicolantonio S, Cipriano F, Pietropaoli D, Ortu E. Trigeminal electrical stimulation with ULFTENS of the dorsal anterior mucosal surface of the tongue: Effects on Heart Rate Variability (HRV). PLoS One. 2023 May 10;18(5):e0285464. doi: 10.1371/journal.pone.0285464. eCollection 2023. PMID 37163499
- [Result] Monaco A, Cattaneo R, Di Nicolantonio S, Strada M, Pietropaoli D, Ortu E. Effects of trigeminal neurostimulation on heart rate variability: comparing cutaneous (Tragus) and tongue (Antero-Dorsal mucosa) stimulation. BMC Oral Health. 2024 Oct 20;24(1):1257. doi: 10.1186/s12903-024-04914-2. PMID 39428464